CLINICAL TRIAL: NCT07078903
Title: Relationship Between Cognitive Impairment and Gait Balance in Chronic Stroke Survivors: A Cross-Sectional Study
Brief Title: Cognitive Impairment and Gait Balance in Chronic Stroke Survivors
Status: Not yet recruiting | Type: Observational
Sponsor: Islam Hassan Fayed (Other)
Collaborators: Majmaah University (Other)
Responsible Party: Sponsor-Investigator, Islam Hassan Fayed, Principal Investigator, Assistan Professor, Cairo University
Organization: Cairo University (Other)
Other Study IDs: MUREC-March.17/COM-2021/30-3
Record Dates: First submitted 2025-07-14; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Chronic Stroke Patients
Keywords: Cognitive Impairment; Chronic Stroke; Gait Balance
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic Stroke Survivors: A group of 26 adults with chronic stroke will be assessed to examine the relationship between cognitive impairment and gait balance. Cognitive function will be evaluated using the Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE), and balance will be assessed using center of pressure measurements with eyes open and closed

SUMMARY:
This study aims to investigate the relationship between cognitive impairment and gait balance in individuals with chronic stroke. Using the IQCODE and a balance assessment system, the study evaluates how post-stroke cognitive decline may influence stability and motor control. The findings will support better rehabilitation strategies tailored to cognitive function.

DETAILED DESCRIPTION:
Cognitive and motor impairments are common consequences of stroke, but they are often treated separately. A growing body of evidence suggests a potential link between cognitive function and physical performance, including balance and gait. This prospective, cross-sectional study investigates the relationship between post-stroke cognitive impairment and gait balance in chronic stroke survivors. Participants will undergo cognitive evaluation using the Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE), and gait balance will be assessed through center of pressure velocity with eyes open and closed. The goal is to identify whether cognitive decline is associated with impaired balance performance and to explore the influence of age, stroke type, and duration on these outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 25-75 years
* Diagnosed with chronic stroke (≥6 months post-stroke)
* Able to stand independently for testing
* Capable of completing assessments or has an informant available for IQCODE

Exclusion Criteria:

* Severe visual, vestibular, or musculoskeletal impairments
* History of other neurological disorders
* Acute illness or uncontrolled medical condition
* Inability to follow instructions or complete cognitive/balance assessments

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A non-random sample of 26 adults aged 25-75 years with chronic stroke, recruited from outpatient rehabilitation centers. Participants were assessed in a single session to evaluate the relationship between cognitive impairment and gait balance.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Correlation between IQCODE scores and center of pressure velocity (eyes open) | At baseline (single session)
  Assess the relationship between cognitive impairment and balance control by comparing IQCODE scores with center of pressure velocity during quiet standing with eyes open.

SECONDARY OUTCOMES:
Correlation between IQCODE scores and center of pressure velocity (eyes closed) | At baseline (single session)
  Assess the relationship between cognitive impairment and postural control by comparing IQCODE scores with center of pressure velocity during quiet standing with eyes closed.

IPD SHARING:
Plan to Share IPD: No
Your dataset is small, with identifiable clinical information, which raises privacy and ethical concerns.
  There's no formal plan in place for anonymized data sharing.
  Most ICMJE-compliant journals accept a "No" or "Undecided" answer, especially for observational studies that do not involve public databases.